CLINICAL TRIAL: NCT02465099
Title: Perioperative Outcomes of Multilevel Posterior Spinal Fusion in Adolescent Scoliosis With Two Energy Dissection Techniques
Brief Title: Posterior Spinal Fusion With Two Energy Dissection Techniques
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated due to commercial considerations with no patient safety reasons.
Sponsor: Ethicon Endo-Surgery (Industry)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENG 14-004
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Electrocautery Dissection (ED) (Active Comparator): Patients meeting the study criteria, scheduled to undergo posterior spinal fusion (PSF) using monopolar electrocautery and metal Cobb elevator (considered the current standard) for soft tissue dissection and removal from vertebral surfaces.
  Interventions: Device: Electrocautery Dissection (ED)
- Ultrasonic Dissection (UD) (Experimental): Patients meeting the study criteria, scheduled to undergo PSF using ultrasonic dissection and metal Cobb elevator for soft tissue dissection and removal from vertebral surfaces.
  Interventions: Device: Ultrasonic Dissection (UD)

INTERVENTIONS:
Device: Ultrasonic Dissection (UD) — Ultrasonic energy will be used as the primary means for soft tissue dissection in patients diagnosed with adolescent scoliosis undergoing multilevel (>=6) PSF
  Other Names: Harmonic ultrasonic dissection
  Arms: Ultrasonic Dissection (UD)
Device: Electrocautery Dissection (ED) — Electrocautery dissection will be used as the primary means for soft tissue dissection in patients diagnosed with adolescent scoliosis undergoing multilevel (>=6) PSF
  Arms: Electrocautery Dissection (ED)

SUMMARY:
The OSTEOVUE™ Spine Dissector is a new ultrasonic energy device, specifically designed for soft tissue removal from vertebral surfaces. The aim of the present study is to compare blood loss in multilevel PSF surgeries in patients with adolescent scoliosis (idiopathic or neuromuscular) done with ED or with UD. Blood loss will be estimated by major intraoperative surgical Stage (1 and 2) and postoperatively (until discharge). Additionally, the study will assess the possible influence of the device use in secondary perioperative outcomes.

DETAILED DESCRIPTION:
The primary objective is to compare intraoperative blood loss between surgeries performed with monopolar electrocautery and ultrasonic energy (as the primary means for soft tissue dissection) in patients diagnosed with adolescent scoliosis undergoing multilevel (>=6) posterior spinal fusion (PSF).

This is a prospective, multicenter, pair-matched comparison study that will be carried out in two phases:

Phase I Perioperative outcome variables (primary and secondary) will be collected from patients with adolescent scoliosis, meeting the study inclusion criteria, scheduled to undergo PSF using monopolar electrocautery and metal Cobb elevator (considered the current standard) for soft tissue dissection and removal from vertebral surfaces. This group will be the Electrocautery Dissection (ED) group.

Phase II The same outcomes variables measured on the ED group during Phase I will be subsequently collected from a group of patients with adolescent scoliosis, meeting the study inclusion criteria and scheduled to undergo PSF surgery. For this study group, surgery will be performed with the Harmonic OSTEOVUE™ Spine Soft Tissue Dissector (referred to as the OSTEOVUE™ Dissector in this protocol) and metal Cobb elevator, as the primary means of soft tissue dissection and removal from vertebral surfaces. This group will be the Ultrasonic Dissection (UD) group.

Patients in the UD group will be recruited from the existing patient population of PSF candidates at each participating site.

Prior to recruitment of participants in Phase II, each Principal Investigator (PI) will have documented training/in service of the use the OSTEOVUE™ Dissector in at least 5 multilevel spine surgery cases.

The proportion of neuromuscular versus idiopathic cases recruited in Phase II will be based on the proportion of patients with either of these conditions recruited in Phase I.

Up to five US sites of orthopedic surgeons and/or neurosurgeons, with expertise in pediatric PSF surgery, will participate in the study. 100 subjects will be enrolled in this study (46 in the ED group and 54 in the UD group).

Propensity score matching will be utilized to match subjects in the ED group to subjects in the UD group. Propensity scores will be based on the variables known to influence blood loss, and full details of the matching methodology will be provided in a separate Statistical Analysis Plan.

ELIGIBILITY:
Inclusion Criteria:

1. Between 10 and 21 years of age;
2. Diagnosed with neuromuscular scoliosis associated with cerebral palsy or with idiopathic scoliosis between the ages of 10 and 18;
3. Indicated for primary PSF surgery;
4. Anticipated >= 6 vertebrae fusions;
5. Not in need of three column osteotomy (pedicle subtraction osteotomy [PSO]);
6. Not in need of vertebral column resection (VCR);
7. Curve magnitude >45 degrees for scoliosis and for sagittal deformity; and
8. An American Society of Anesthesiologists (ASA) physical status (PS) classification of 1 to 4

Exclusion Criteria:

1. One or both parents or a guardian unable or unwilling to provide parental permission and child assent (if capable, the child must express willingness to participate);
2. Previous failed vertebral fusion at same target levels;
3. Syndromic scoliosis;
4. Congenital scoliosis;
5. Early-onset scoliosis (onset before 10 years of age);
6. Requiring an anterior procedure;
7. Requiring PSO;
8. Requiring VCR;
9. Presence of coagulation abnormalities;
10. Planned staged procedure (exclude if second stage or beyond);
11. Requiring emergency surgery; and/or
12. Participation in any other clinical study (not to include registry or survey-only studies) for the duration of the study.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2016-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Kassis, M.D., Study Director — Ethicon, Inc.
Locations (5):
- United States (5):
  - Valley Children's Hospital, Madera, California
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Shriners Hospital for Children - Chicago, Chicago, Illinois
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Shriners Hospitals for Children-Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available.

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Monopolar Electrocautery Dissection: Patients meeting the study criteria, scheduled to undergo posterior spinal fusion using monopolar electrocautery and metal Cobb elevator (considered the current standard) for soft tissue dissection and removal from vertebral surfaces.
- Phase II OSTEOVUE Ultrasonic Dissection: Patients meeting the study criteria, scheduled to undergo posterior spinal fusion using ultrasonic dissection and metal Cobb elevator for soft tissue dissection and removal from vertebral surfaces.
Period: Overall Study
Arm/Group | Phase 1 Monopolar Electrocautery Dissection | Phase II OSTEOVUE Ultrasonic Dissection
Started | 45 | 19
Completed | 45 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Monopolar Electrocautery Dissection | Phase II OSTEOVUE Ultrasonic Dissection | Total
Number analyzed (Participants) | 45 | 19 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.1 (2.64) | 14.5 (1.84) | 14.9 (2.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 14 | 51
  Male | 8 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 31 | 16 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 45 | 19 | 64

OUTCOME MEASURES:

1. Primary Outcome: Estimated Intraoperative Blood Loss
Description: Estimated blood loss during intraoperative Stage 1, defined as the period from first incision to the first bone violation/cut (e.g., first pedicle screw drill); and intraoperative Stage 2, defined as the period from first bone violation/cut to last suture.
Time Frame: Intraoperative
Population: All subjects in which the procedure was started. There was one subject that was enrolled who was to receive treatment with ultrasonic dissection, but the procedure was not performed due to study closure. Therefore, N=19 subjects enrolled for the ultrasonic dissection group, but only 18 subjects received treatment.
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Phase 1 Monopolar Electrocautery Dissection | Phase II OSTEOVUE Ultrasonic Dissection
Number analyzed (Participants) | 45 | 18
milliliters | 134 (124) | 163 (146)

ADVERSE EVENTS:
Time Frame: Intraoperatively through hospital discharge (average of 5 days with range of 2 to 24 days).
Description: All AEs attributable to the use of monopolar electrocautery dissection or OSTEOVUE ultrasonic dissection devices were recorded. Postop bleeding resulting in hospital readmission/reop was considered a reportable AE irrespective of relationship to either study device. One subject was enrolled to receive treatment with ultrasonic dissection, but the procedure was not performed due to study closure. N=19 subjects enrolled for the ultrasonic dissection group, but only 18 subjects received treatment.
Arm/Group | Phase 1 Monopolar Electrocautery Dissection | Phase II OSTEOVUE Ultrasonic Dissection
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/18
Other Adverse Events (participants affected / at risk) | 0/45 | 0/18

LIMITATIONS AND CAVEATS:
Study was terminated due to internal strategic considerations and not for any patient safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed that the first publication of results should be made in conjunction with the presentation of a joint, multicenter publication of the results with all sites contributing data, analyses, and comments. If this publication was not submitted within 12 months after conclusion of the Study at all sites, or after Sponsor confirmed there would be no multicenter Study publication, whichever is first, the PIs could have published the results from their individual sites.